CLINICAL TRIAL: NCT00375284
Title: A Phase IV Randomised, Double-blind, Active and Placebo-controlled, 6-week Trial to Investigate the Efficacy and Safety of a Starting (and Fixed) Dose 0.25 mg Pramipexole (Mirapex®) in Patients With Idiopathic Restless Legs Syndrome
Brief Title: A 6 Week Trial to Study the Efficacy and Safety of a Starting Dose 0.25 mg Pramipexole (Mirapex) in Patients With RLS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 248.616
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Pramipexole

INTERVENTIONS:
Drug: Pramipexole

SUMMARY:
This trial is a 6-week, double-blind, randomized, active and placebo-controlled parallel-group study with a primary objective of comparison of starting doses of pramipexole fixed-dose (0.25 mg daily) and pramipexole titrated-dose (0.125 mg qd for 1 week, then 0.25 mg qd for the remaining 5 weeks) with placebo to evaluate efficacy and safety in treating RLS symptoms in patients diagnosed with idiopathic RLS.

The secondary objectives of this study will be to assess the onset of action of symptomatic relief of RLS for pramipexole with daily assessment of PGI and modified IRLS during two intervals of the first 2 weeks (Days 2, 3 and 4 and Days 9, 10, and 11) and assessment of IRLS, PGI and CGI-I at Weeks 1, 2, 4 and 6 (CGI-I additionally on Day 3).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent consistent with ICH-GCP and local IRB/IEC requirements obtained prior to any study procedures being performed and the ability and willingness to comply with study treatment regimen and to attend study assessments.
2. Male or female out-patients 18 to 80 years of age.
3. Diagnosis of idiopathic RLS according to the clinical RLS criteria revised by the IRLSSG in collaboration with the U.S.A. National Institutes of Health [P03-03355]. All four criteria must be present to fulfil the diagnosis of RLS:

   - An urge to move the legs, usually accompanied or caused by uncomfortable and unpleasant sensations in the legs. (Sometimes the urge to move is present without the uncomfortable sensations and sometimes the arms or other body parts are involved in addition to the legs).

   The urge to move or unpleasant sensations begin or worsen during periods of rest or inactivity such as lying or sitting.
   * The urge to move or unpleasant sensations are partially or totally relieved by movement, such as walking or stretching, at least as long as the activity continues.
   * The urge to move or unpleasant sensations are worse in the evening or night than during the day or only occur in the evening or night. (When symptoms are very severe, the worsening at night may not be noticeable but must have been previously present).
4. RLS symptoms present at least 2 to 3 days per week during the last 3 months.
5. IRLS rating scale score >15 at baseline (Visit 2).

Exclusion Criteria:

1. Women of child-bearing potential (i.e., premenopausal women, or postmenopausal women less than 6 months after last menses) who do not use during the clinical trial an adequate method of contraception such as: double barrier protection (e.g., diaphragm or condom and spermicide), intrauterine device, hormonal therapy (oral, injectable, or subcutaneous), or partners surgical sterilization.
2. Any women of child-bearing potential not having negative pregnancy test at screening.
3. Breastfeeding women.
4. Concomitant or previous pharmacologic therapy for RLS as follows:

   * Any intake of dopamine agonists within 14 days prior to baseline (Visit 2).
   * Any intake of L-dopa within 14 days prior to baseline (Visit 2).
   * Any intake of L-dopa prior to baseline visit, if augmentation in RLS symptoms was observed.
   * Unsuccessful prior treatment with non-ergot dopamine agonists (e.g., pramipexole, ropinirole).
5. All treatment less than 14 days before baseline (Visit 2) or concomitant treatment with medication or dietary supplements which could significantly influence RLS symptoms, e.g., dopaminergic (other than levodopa and dopamine agonists) or antidopaminergic drugs, non-selective MAO inhibitors, sympathomimetics, neuroleptics, antidepressants, hypnotics, any benzodiazepines, antiepileptics, opioids, clonidine, ferrous salts, magnesium, folic acid, vitamin B12, antihistaminics, lithium, metoclopramide.
6. Withdrawal symptoms of any medication must not be present at baseline (Visit 2).
7. Previous pramipexole non-responders in other indications than RLS.
8. Patients with known hypersensitivity to pramipexole or any other component of the investigational product or placebo tablets.
9. Confirmed diagnosis of diabetes mellitus requiring insulin therapy.
10. Any of the following lab results at screening:

    * Patients with any clinically significant abnormalities in laboratory parameters at screening at the investigators discretion.
    * Haemoglobin (Hb) below lower limit of normal (LLN).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2006-09; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The co-primary endpoints are: Assessment of clinical response of treatment measured by the change from baseline in total IRLS score and CGI-I responder rate (at least much improved) after 6 weeks, 2 weeks and 1 week. | 6 weeks

SECONDARY OUTCOMES:
Onset of action on Day 3 as measured by the CGI-I responder rate Onset of action as measured by PGI and modified IRLS score Clinical Global Impression of improvement Patient Global Impression IRLS as a responder rate VAS score for pain in limbs | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (52):
- United States (52):
  - 248.616.065 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 248.616.028 Boehringer Ingelheim Investigational Site, Dothan, Alabama
  - 248.616.035 Boehringer Ingelheim Investigational Site, Mesa, Arizona
  - 248.616.025 Boehringer Ingelheim Investigational Site, Peoria, Arizona
  - 248.616.073 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 248.616.067 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 248.616.009 Boehringer Ingelheim Investigational Site, Fayetteville, Arkansas
  - 248.616.040 Boehringer Ingelheim Investigational Site, Foothill Ranch, California
  - 248.616.062 Boehringer Ingelheim Investigational Site, Fullerton, California
  - 248.616.050 Boehringer Ingelheim Investigational Site, Pasadena, California
  - 248.616.031 Boehringer Ingelheim Investigational Site, Colorado Springs, Colorado
  - 248.616.017 Boehringer Ingelheim Investigational Site, Pueblo, Colorado
  - 248.616.071 Boehringer Ingelheim Investigational Site, Wallingford, Connecticut
  - 248.616.043 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 248.616.014 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 248.616.020 Boehringer Ingelheim Investigational Site, Naples, Florida
  - 248.616.048 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 248.616.072 Boehringer Ingelheim Investigational Site, Spring Hill, Florida
  - 248.616.018 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 248.616.049 Boehringer Ingelheim Investigational Site, Augusta, Georgia
  - 248.616.033 Boehringer Ingelheim Investigational Site, Columbus, Georgia
  - 248.616.057 Boehringer Ingelheim Investigational Site, Macon, Georgia
  - 248.616.066 Boehringer Ingelheim Investigational Site, Savannah, Georgia
  - 248.616.047 Boehringer Ingelheim Investigational Site, Stockbridge, Georgia
  - 248.616.059 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 248.616.045 Boehringer Ingelheim Investigational Site, Lenexa, Kansas
  - 248.616.061 Boehringer Ingelheim Investigational Site, Olathe, Kansas
  - 248.616.060 Boehringer Ingelheim Investigational Site, Baton Rouge, Louisiana
  - 248.616.058 Boehringer Ingelheim Investigational Site, Brighton, Massachusetts
  - 248.616.051 Boehringer Ingelheim Investigational Site, Wellesley Hills, Massachusetts
  - 248.616.001 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 248.616.004 Boehringer Ingelheim Investigational Site, Jackson, Mississippi
  - 248.616.064 Boehringer Ingelheim Investigational Site, Florissant, Missouri
  - 248.616.016 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 248.616.063 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 248.616.053 Boehringer Ingelheim Investigational Site, Dover, New Hampshire
  - 248.616.036 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 248.616.021 Boehringer Ingelheim Investigational Site, Albany, New York
  - 248.616.013 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 248.616.003 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 248.616.068 Boehringer Ingelheim Investigational Site, Marion, Ohio
  - 248.616.012 Boehringer Ingelheim Investigational Site, Norman, Oklahoma
  - 248.616.006 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 248.616.019 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 248.616.069 Boehringer Ingelheim Investigational Site, Clarks Summit, Pennsylvania
  - 248.616.008 Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - 248.616.005 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 248.616.070 Boehringer Ingelheim Investigational Site, Rockwall, Texas
  - 248.616.039 Boehringer Ingelheim Investigational Site, San Marcos, Texas
  - 248.616.011 Boehringer Ingelheim Investigational Site, Alexandria, Virginia
  - 248.616.055 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - 248.616.024 Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin